CLINICAL TRIAL: NCT05404048
Title: Programmed Death Ligand 1 (PD-L1)-PET Imaging in Patients With (Diffuse) Large B-cell Lymphoma Who Are Treated With CD19-directed CAR T-cell Therapy: a Pilot Study
Brief Title: PD-L1 PET-imaging During CAR T-cell Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202100663
Record Dates: First submitted 2022-05-05; First posted 2022-06-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Large B-cell Lymphoma
Keywords: PD-L1; CAR T-cell therapy; Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-L1 PET-imaging (Experimental): The main intervention of this study is 89Zr-atezolizumab PET-scan combined with a low-dose CT-scan. The PET/CT scan will be performed before infusion of CAR T-cell therapy. In patients with an end-of-treatment F-FDG positive PET-signal a second 89Zr-atezolizumab PET/CT-scan will be performed.
  Interventions: Other: 89Zr-atezolizumab PET-imaging

INTERVENTIONS:
Other: 89Zr-atezolizumab PET-imaging — 89Zr-atezolizumab tracer injection + PET/CT-scan

SUMMARY:
This is a single-center, single-arm pilot trial designed to evaluate the expression of PD-L1 in patients with Large B-cell lymphoma (LBCL) and its role in non-responsiveness to chimeric antigen receptor (CAR) T-cell therapy in a non-invasive manner. Moreover, within this trial 89Zr-atezolizumab PET/CT imaging as a tool to distinguish lymphoma activity from a treatment-related inflammatory signal (histiocytic/sarcoid-like reaction) in patients with an end-of-treatment positive FDG PET/CT signal will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed LBCL and associated subtypes, defined by WHO 2016 classification
* Tumor lesion(s) of which a histological biopsy can safely be obtained according to Standard clinical care procedures.
* Measurable disease, as defined by Lugano criteria.
* If has history of central nervous system (CNS) disease, then must have no signs or symptoms of CNS disease, no active disease on magnetic resonance imaging (MRI) and absence of large cell lymphoma in cerebral spinal fluid (CSF) on cytospin preparation and flow cytometry, regardless of the number of white blood cells.
* If has history of cerebral vascular accident (CVA), the CVA event must be 12 months prior to apheresis and any neurological deficits must be stable.
* Signed informed consent.
* Age >18 at the time of signing informed consent.
* Life expectancy >12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Ability to comply with the protocol.

Exclusion Criteria:

* Signs or symptoms of active infection within 2 weeks prior to 89Zr-atezolizumab injection, unless treated to resolution.
* Prior CD19-directed CAR T-cell therapy or other bi-specific antibodies targeting CD19 receptor (e.g.blinatumomab).
* History of severe allergy, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of 89Zr-atezolizumab, or that may affect the interpretation of the results or render the patient at high risk for complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
To evaluate the expression of PD-L1 in normal tissue and lymphoma lesions before CAR T-cell therapy by 89Zr-atezolizumab PET/CT imaging. | 2 year
To correlate the pretreatment 89Zr-atezolizumab uptake to the objective response rate to CAR T-cell therapy. | 2 year
To evaluate the utility of the 89Zr-atezolizumab uptake to distinguish lymphoma activity from a treatment-related inflammatory reaction in patients with an end-of-treatment 18F-FDG-positive PET/CT signal. | 2 year

SECONDARY OUTCOMES:
To correlate the pretreatment 89Zr-atezolizumab distribution to CAR T-cell peak expansion and persistence. | 2 year
To correlate the pretreatment 89Zr-atezolizumab uptake to CAR T-cell therapy related grade 1-5 adverse events (cytokine release syndrome (CRS) and immune effector cell associated neurotoxicity syndrome (ICANS)). | 2 year
To correlate tumor 89Zr-atezolizumab uptake with tumor and immune cell PD-L1 expression as assessed by immunohistochemistry on a fresh contemporaneous tumor biopsy. | 2 year
To compare the 89Zr-atezolizumab distribution in irradiated versus non-irradiated lymphoma lesions in patients who require radiotherapy as a bridging strategy prior to CAR T-cell infusion. | 2 year
To determine the incidence of a treatment-related inflammatory signal on 18F-FDGPET/CT scan (histiocytic/sarcoid-like reaction) after CAR T-cell therapy. | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Tom van Meerten, MD,PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT05404048/Prot_SAP_000.pdf